CLINICAL TRIAL: NCT05752500
Title: Optimization of a Behavioral Intervention to Increase Physical Activity in Older Adults Living With HIV
Acronym: HiActivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2208-002
Record Dates: First submitted 2023-02-22; First posted 2023-03-02 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Hiv; Physical Inactivity; Aging
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sedentary Behavior | interventions — Exercise; Crisis Intervention

STUDY DESIGN:
Intervention Model Description: 2x2x2 factorial design
Who Masked: Investigator
Masking Description: Data analyst will be masked to intervention component assignment labels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- BASM + PA Coaching (Experimental): Brief Advice and Self-Monitoring Physical Activity Coaching
  Interventions: Behavioral: Physical Activity Coaching; Behavioral: Brief Advice and Self-Monitoring
- BASM + CB-PA (Experimental): Brief Advice and Self-Monitoring Cognitive-Behavioral Intervention to Increase Physical Activity
  Interventions: Behavioral: Cognitive Behavioral Intervention for Physical Activity; Behavioral: Brief Advice and Self-Monitoring
- BASM + SS-PA (Experimental): Brief Advice and Self-Monitoring Social support for Physical Activity
  Interventions: Behavioral: Social Support for Physical Activity; Behavioral: Brief Advice and Self-Monitoring
- BASM + PA Coaching + CB-PA (Experimental): Brief Advice and Self-Monitoring Physical Activity Coaching Cognitive-Behavioral Intervention to Increase Physical Activity
  Interventions: Behavioral: Cognitive Behavioral Intervention for Physical Activity; Behavioral: Physical Activity Coaching; Behavioral: Brief Advice and Self-Monitoring
- BASM + PA Coaching + SS-PA (Experimental): Brief Advice and Self-Monitoring Physical Activity Coaching Social support for Physical Activity
  Interventions: Behavioral: Social Support for Physical Activity; Behavioral: Physical Activity Coaching; Behavioral: Brief Advice and Self-Monitoring
- BASM + CB-PA + SS-PA (Experimental): Brief Advice and Self-Monitoring Cognitive-Behavioral Intervention to Increase Physical Activity Social support for Physical Activity
  Interventions: Behavioral: Cognitive Behavioral Intervention for Physical Activity; Behavioral: Social Support for Physical Activity; Behavioral: Brief Advice and Self-Monitoring
- BASM + PA Coaching + CB-PA + SS-PA (Experimental): Brief Advice and Self-Monitoring Physical Activity Coaching Cognitive-Behavioral Intervention to Increase Physical Activity Social support for Physical Activity
  Interventions: Behavioral: Cognitive Behavioral Intervention for Physical Activity; Behavioral: Social Support for Physical Activity; Behavioral: Physical Activity Coaching; Behavioral: Brief Advice and Self-Monitoring
- BASM (Other): Brief Advice and Self-Monitoring
  Interventions: Behavioral: Brief Advice and Self-Monitoring

INTERVENTIONS:
Behavioral: Cognitive Behavioral Intervention for Physical Activity — Interventionist will use cognitive and behavioral techniques to help the participant increase facilitators and decrease barriers to physical activity, particularly barriers such as lack of motivation, depression, and chronic pain. Meetings will occur every other week for 4 months.
  Other Names: CB- PA
  Arms: BASM + CB-PA; BASM + CB-PA + SS-PA; BASM + PA Coaching + CB-PA; BASM + PA Coaching + CB-PA + SS-PA
Behavioral: Social Support for Physical Activity — This component will leverage the social functionality of the Fitbit app, promoting social support and friendly competition via a moderated Facebook group.
  Other Names: SS-PA
  Arms: BASM + CB-PA + SS-PA; BASM + PA Coaching + CB-PA + SS-PA; BASM + PA Coaching + SS-PA; BASM + SS-PA
Behavioral: Physical Activity Coaching — The PA coach will meet with the participant to set goals for physical activity (steps) and encourage self-monitoring. Meetings will occur every other week for 4 months.
  Other Names: PA Coaching
  Arms: BASM + PA Coaching; BASM + PA Coaching + CB-PA; BASM + PA Coaching + CB-PA + SS-PA; BASM + PA Coaching + SS-PA
Behavioral: Brief Advice and Self-Monitoring — Participants will receive a single session with brief advice about increasing physical activity, and instructions on how to use their study-provided FitBit.
  Other Names: BASM

SUMMARY:
The goal of this clinical trial is to examine 3 interventions designed to increase physical activity in older adults with HIV. We will examine 3 potential components of an intervention package: physical activity coaching, cognitive behavioral therapy targeted toward common barriers to physical activity such as low motivation or chronic pain, and a Fitbit-based social support intervention. Our primary outcome will be physical activity, defined as steps per day. Results will guide choice of intervention components to be used in an optimized behavioral intervention.

DETAILED DESCRIPTION:
Increasing numbers of persons living with HIV (PLWH) are living to older ages. Older PLWH are at increased risk for a wide spectrum of co-morbid conditions such as cardiovascular disease, frailty phenotype, and mental health disorders. Practical primary care-based interventions are needed for older PLWH that target lifestyle factors to reduce complications of aging and improve healthspan. Most PLWH engage in less physical activity (PA) than is recommended by public health guidelines. Thus, increasing PA can lead to numerous mental and physical health benefits among PLWH. Current studies in PLWH typically focus on the impact of supervised exercise. However, there are many barriers to this type of PA. Lifestyle physical activity (LPA) programs that focus on integrating PA, especially walking, into everyday life, may be more successful in producing a sustained increase in PA. The long-term goal of this research is to develop an effective and efficient primary care intervention that increases LPA among older PLWH. We leverage the Multiphase Optimization STrategy (MOST) as a framework for developing, optimizing, and evaluating a multicomponent behavioral intervention. MOST is comprised of three phases. First, in the preparation phase, an empirical and theory-driven conceptual model is developed that identifies differentiable intervention components and specifies optimization criteria (i.e., goal of intervention development). We have completed this phase. Second, in the optimization phase, the impact of each intervention component on the desired outcome is empirically examined. The goal is to determine which components to include in a final intervention package that is optimized for efficacy and efficiency. The proposed study reflects the second phase, or an optimization trial. Finally, in the evaluation phase, the optimized intervention package is evaluated for efficacy in a traditional RCT; this will be the next step in this line of research following the currently proposed project. In this project, we will test the impact of three separable intervention components on steps per day after 4 months of intervention. We will recruit 208 PLWH of age ≥50 year classified as low-active. All participants receive component '0': brief advice to exercise and a Fitbit activity tracker. We then test 3 additional components in a factorial design: 1) PA Coaching-focused on goal-setting and self-monitoring; 2) Cognitive-Behavioral intervention for PA (CB-PA)-focused on identifying values and addressing internal barriers to PA such as pain, depression, or fatigue; 3) Social Support for PA (SS-PA)-a component which leverages the social functionality of the Fitbit app, promoting social support and friendly competition. The primary outcome will be steps per day during Month 4. The observed main and interaction effects for the 3 candidate components will guide selection of components to be included in an optimized intervention that will be tested in a future RCT. We will also examine potential mediators for each intervention component, as well as secondary outcomes including perceived physical health, mental health, cardiovascular disease risk, and the frailty phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. HIV positive: defined by HIV antibody, detectable HIV RNA in plasma, or a note from the participant's HIV care provider.
2. Must be on continuous antiretroviral therapy (ART) for > 3 months, as assessed via self-report.
3. Low PA: defined as self-report of < 90 minutes of moderate-vigorous PA (MVPA) per week in the previous 3 months AND less than 14 hours per week of sustained walking in the previous 4 weeks.
4. Medically cleared for moderate PA. If participants report a) a history of cardiovascular disease including known coronary artery disease, peripheral vascular disease, heart failure, or stroke; or b) chest pain, shortness of breath, or dizziness or syncope either at rest or during activity in the past 3 months, then they must have medical clearance by a physician or primary care provider.
5. Age 50 years or older.
6. Proficiency in English: sufficient to engage in informed consent, understand assessments and materials provided, and engage and use Fitbit application (all materials provided in English).
7. Capacity to consent, documented by acceptable answers in a consent "teach-back" process.
8. Score of greater than 16 on the MOCA
9. Able to ambulate without assistive devices
10. Ability to use the FitBit application, as demonstrated to study staff.

Exclusion Criteria:

* Exclusion Criteria

  1. Medical conditions or physical or neurocognitive limitations that interfere with PA or study participation.
  2. Hazardous substance use, assessed via a score ≥15 on the Alcohol Use Disorders Identification Test (AUDIT) or ≥6 on the Drug Abuse Screening Test (DAST).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Steps per day | Month 4
  Assessed via Fitbit

SECONDARY OUTCOMES:
Minutes per week of moderate-vigorous activity | Month 4
  Assessed via FitBit
Minutes per week of moderate-vigorous activity, self-report | Month 4
  Assessed via the International Physical Activity Questionnaire
Frailty Phenotype | Month 4
  Assessed via the Fried Criteria
CVD Risk | Month 4
  Assessed using Life's Simple 7 Scale
Physical performance | Month 4
  Assessed via the Short Physical Performance Battery
Emotional Well-being | Month 4
  Assessed via PROMIS-29 v2.1 profile - Mental Health summary score
Physical functioning | Month 4
  Assessed via PROMIS-29 v2.1 profile - Physical Health summary score

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Uebelacker, PhD, Principal Investigator — Butler Hospital; Jason Baker, MD, Principal Investigator — Hennepin Healthcare
Locations (2):
- United States (2):
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - Lifespan Affiliates, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No